CLINICAL TRIAL: NCT07294898
Title: A Phase 1, Open-Label, Randomized, Crossover Study to Evaluate the Effect of a Low-Fat Meal and Evening Dosing on the Pharmacokinetics of KAI-7535 in Healthy Participants Living With Obesity or Overweight
Brief Title: A Study to Investigate the Effect of a Low-fat Meal and Evening Dosing on KAI-7535 in Participants Living With Obesity or Overweight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kailera (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: K7535-1709
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
Keywords: Obesity; Overweight; Glucagon-like peptide-1; GLP-1; KAI-7535
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- KAI-7535: Morning Dosing, Fed (Experimental): Participants will receive KAI-7535 in the morning following a meal on dosing days.
  Interventions: Drug: KAI-7535
- KAI-7535: Morning Dosing, Fasted (Experimental): Participants will receive KAI-7535 in the morning following an overnight fast on dosing days.
  Interventions: Drug: KAI-7535
- KAI-7535: Evening Dosing (Experimental): Participants will receive KAI-7535 in the evening on dosing days.
  Interventions: Drug: KAI-7535

INTERVENTIONS:
Drug: KAI-7535 — Oral tablets.

SUMMARY:
The primary objective of this study is to evaluate the effect of a meal and evening dosing on the pharmacokinetics (PK) of KAI 7535 in healthy participants living with obesity or overweight.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) ≥25.0 and ≤40.0 kg/m^2.
* Medically healthy, as determined by prestudy medical history, and without clinically significant (CS) abnormalities.

Key Exclusion Criteria:

* Known hypersensitivity to study treatment or any study treatment ingredients.
* History or presence of CS cardiovascular, pulmonary, hepatic, renal, hematological, GI, endocrine, immunologic, dermatologic, psychiatric, or neurological disease/disorder, including any acute illness, within the past 3 months.

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-01-26 (Actual); Study Completion 2026-01-26 (Actual)

PRIMARY OUTCOMES:
Time to Maximum Observed Concentration (Tmax) of KAI-7535 | Pre-dose and up to 60 hours post-dose
Maximum Observed Concentration (Cmax) of KAI-7535 | Pre-dose and up to 60 hours post-dose
Area Under the Concentration-time Curve From 0 to Time of Last Quantifiable Concentration (AUC0-t) of KAI-7535 | Pre-dose and up to 60 hours post-dose
Area Under the Concentration-time Curve From 0 to Infinity (AUC0-inf) of KAI-7535 | Pre-dose and up to 60 hours post-dose

SECONDARY OUTCOMES:
Number of Participants with a Treatment-emergent Adverse Event (TEAE) | Day 1 up to Day 12

CONTACTS AND LOCATIONS:
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No